CLINICAL TRIAL: NCT06277622
Title: A Prospective Multicenter Cohort Study About Internal Fixation Using Proximal Femoral Universal Nail (PFUN) Versus Proximal Femoral Nail Antirotation (PFNA) for Femoral Intertrochanteric Fracture
Brief Title: A Prospective Multicenter Cohort Study About Internal Fixation Using PFUN Versus PFNA for Femoral Intertrochanteric Fracture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Collaborators: Beijing Yanqing Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PekingUTH ZFCY PFUN
Record Dates: First submitted 2024-02-19; First posted 2024-02-26 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-01

CONDITIONS: Femoral Intertrochanteric Fractures
Keywords: Femoral Intertrochanteric Fractures; internal fixation; PFUN and PFNA; multicenter randomized controlled clinical trial; internal fixation failure rate

STUDY DESIGN:
Intervention Model Description: This prospective multicenter cohort study is to compare the post-operative implant failure rate between the patients with femoral intertrochanteric fracture (AO classification 31-A) using Proximal Femoral Universal Nail (PFUN) versus Proximal Femoral Nail Antirotation (PFNA) at 21-month follow up.The patients are divided into the PFUN group and the PFNA group according to the internal fixation they choose.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Proximal Femoral Universal Nail (PFUN) (Experimental)
  Interventions: Device: PFUN
- Proximal Femoral Nail Antirotation (PFNA) (Active Comparator)
  Interventions: Device: PFNA

INTERVENTIONS:
Device: PFUN — perform preoperative preparation, intraoperative operation and internal fixation implantation according to the instructions provided in the product packaging.
  Arms: Proximal Femoral Universal Nail (PFUN)
Device: PFNA — perform preoperative preparation, intraoperative operation and internal fixation implantation according to the instructions provided in the product packaging.
  Arms: Proximal Femoral Nail Antirotation (PFNA)

SUMMARY:
This prospective multicenter cohort study is to compare the post-operative implant failure rate between the patients with femoral intertrochanteric fracture (AO classification 31-A) using Proximal Femoral Universal Nail (PFUN) versus Proximal Femoral Nail Antirotation (PFNA) at 21-month follow up. The patients are divided into the PFUN group and the PFNA group according to the internal fixation they choose. The internal fixation failure rate (IFFR) and differences in fracture prognosis of the two groups will be compared. Obtain clinical data of PFUN in the Chinese population, and verify the safety and efficacy of PFUN for patients with femoral intertrochanteric fracture.

DETAILED DESCRIPTION:
This is a prospective multicenter cohort study. The team leader is Peking University Third Hospital. All patients are divided into 2 groups according to the internal fixation they choose. Investigators use PFUN for internal fixation in Group 1 and PFNA in Group 2. The relevant parameters of the sample calculation are α = 0.05 (one-sided) and β = 0.2. PASS 15 was used for calculation, and the final sample size was 130. The PFUN group and the PFNA group each included 65 patients. See the text for detailed inclusion and exclusion criteria. Patients that meet all the inclusion criteria but do not meet any exclusion criteria, and who have signed the informed consent will be recruited, and each patient will be assigned a unique patient identification number, which will be used throughout the study identify the patient. Investigators will perform preoperative preparation, intraoperative operation and internal fixation implantation according to the instructions provided in the product packaging. Investigators only plan to include cases that can successfully conduct closed reduction, therefore investigators will exclude cases that require open reduction. After the operation, the patients will be managed according to the standard nursing and rehabilitation procedures of the experimental site and the results of laboratory tests will be recorded. Regular follow-up evaluation will be performed after the operation until the end of the 21-month follow-up or the primary end point of the study. In this study, the internal fixation failure rate (IFFR) is used as the primary end point of the study, which is defined as the total incidence of internal plant cut-out and fracture. The results of the radiographic examination, the lateral X-ray film and computed tomography(CT), will be evaluated by an independent radiologist to determine whether there are cut-out or fracture of the internal plant. Secondary endpoints include: 1. Bone nonunion after 36 weeks: evaluate bone healing according to the lateral X-ray examination. According to the regulations of Food and Drug Administration of the US, it is defined as nonunion if there are no obvious signs of fracture healing 9 months after the fracture, or if there is no obvious difference in fracture space after three consecutive months. 2. Garden classification proportion, and Garden index for reduction assessment. 3. Clinical prognosis: o A 12-Item Short-Form Health Survey (SF-12) o Harris hip score. 4. Operation time, from the incision to internal fixation implanted. 5. The times of intraoperative fluoroscopy, average 25 milliseconds per Xray shot, record the number of X-ray shot. 6. Postoperative adverse events within 2 years, including ipsilateral femoral head avascular necrosis, infection, wound hematoma, ipsilateral coxa vara, and ipsilateral limb shortening. In this study, it is difficult to blind anyone . Investigators will try their best to reduce human-induced bias in experimental results. Investigators will use one-sided α = 0.05 for statistical tests and confidence interval calculations. P value <0.05 is considered statistically significant. SPSS (latest version: SPSS Inc., Chicago, IL, USA) will be used to analyze the results

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Patients with unilateral femoral intertrochanteric fractures that will be treated with internal fixation
3. According to AO fracture classification, subjects with the fracture type (31-A)
4. Subjects (with the help of relatives) can understand the informed documents and patient questionnaires.
5. Subjects (with the help of relatives) voluntarily provide written informed consent to participate in the clinical study and authorize the transfer of their information to the sponsor.
6. The investigator believes that the subject can understand the clinical study, is willing and able to complete all research procedures and followup visits and can cooperate with the research procedures.
7. In-label use of the PFUN and PFNA.

Exclusion Criteria:

1. Subject does not provide voluntary consent to participate in the study.
2. The researcher believes that the subjects have conditions that affect the participation and follow-up of this study. (for example, the patient lives in a remote area or has difficulty in going back to the hospital for follow-up or does not cooperate with the medical guidance and suggestions of the surgeon.)
3. The subjects were pregnant or lactating women.
4. The researchers believe that the subjects have psychological disorders, which may affect the treatment outcome.
5. Subjects have significant neurological or musculoskeletal disorders or may have adverse effects on gait or weight-bearing (e.g., muscular dystrophy, multiple sclerosis, cerebral infarction, hemiplegia, Charcot arthropathy, avascular necrosis of the femoral head).
6. Concurrent hip osteoarthritis.
7. Fractures where the operative treatment will occur more than three weeks after the primary injury
8. Patients combined with other bone fractures.
9. Pathological fracture (e.g., primary or metastatic tumor)
10. Serious soft tissue injury, judged by the investigator, will impact the union of the fracture, combined open fractures, vascular injury, and combined osteofascial compartment syndrome
11. Multiple systemic injuries judged by researchers not suitable for enrollment.
12. Revision surgeries (for example, due to malunion, nonunion or infection)
13. Concurrent medical conditions judged by researchers not suitable for enrollment, such as: metabolic bone disease, post-polio syndrome, poor bone quality, prior history of poor fracture healing, etc
14. Patients with anaesthetic and surgical contraindications
15. Patients known to be allergic to implant components
16. Patients who are currently using chemotherapeutics or accepting radiotherapy, use systematically corticosteroid hormone or growth factor, or long-term use sedative hypnotics (continuous use over 3 months) or non-steroidal anti-inflammatory drugs (continuous use over 3 months)
17. Intemperance judged by researchers not suitable for enrollment (e.g., excessive daily drinking or smoking, drug abuse);
18. Subjects participated in other clinical studies in the past 3 months, which may affect the outcome and follow-up according to the judgment of researchers.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Internal fixation failure rate | from operation to 21-month follow-up after the surgery
  defined as the total incidence of internal plant cut-out and fracture.

SECONDARY OUTCOMES:
Number of Participants with Bone nonunion | from operation to 21-month follow-up after the surgery
  evaluate bone healing according to the lateral X-ray examination. According to the regulations of Food and Drug Administration of the US, if there are no obvious signs of fracture healing 9 months after the fracture, or if there is no obvious difference in fracture space after three consecutive months, it is defined as nonunion.
Harris hip score | from operation to 21-month follow-up after the surgery
  the score value is from 0 to 100, and a higher score means a better outcome
operation time | intraoperative
  from the incision to internal fixation implanted.
The times of intraoperative fluoroscopy | intraoperative
  average 25 milliseconds per X-ray shot, record the number of X-ray shot
Number of Participants with Postoperative adverse events | from operation to 21-month follow-up after the surgery
  including ipsilateral femoral head avascular necrosis, infection, wound hematoma, ipsilateral coxa vara, and ipsilateral limb shortening

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No